CLINICAL TRIAL: NCT01271231
Title: Effects of Periodontal Treatment on Clinical Parameters and Glucose Metabolism in Diabetic Patients
Brief Title: Study on Periodontal Treatment in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Principal Investigator, Javier Enrique Botero, Assistant Professor, Universidad de Antioquia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 020-2009
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes; Gingivitis; Periodontitis
Keywords: periodontal treatment, diabetes, glycemia, glycated hemoglobin
MeSH Terms: conditions — Diabetes Mellitus; Gingivitis; Periodontitis | interventions — Tooth Exfoliation; Root Planing; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Group IP1 (Placebo Comparator)
  Interventions: Drug: Scaling and root planing plus placebo
- Group IP2 (Experimental)
  Interventions: Drug: Scaling and root planing plus azythromycin
- Group IP3 (Active Comparator)
  Interventions: Drug: Prophylaxis plus azythromycin

INTERVENTIONS:
Drug: Scaling and root planing plus placebo — Single session of scaling and root planing using ultrasonic device. placebo tablets 500 mg, 1 tablet every 24 hours for 3 days
  Arms: Group IP1
Drug: Scaling and root planing plus azythromycin — Single session of scaling and root planing using ultrasonic device. Azythromycin tablets 500mg. 1 tablet every 24 hours for 3 days.
  Arms: Group IP2
Drug: Prophylaxis plus azythromycin — Dental polishing using prophylaxis paste and rubber cups. Azythromycin tablets 500mg. 1 tablet every 24 hours for 3 days.
  Arms: Group IP3

SUMMARY:
Diabetes is a metabolic disorder that affects the uptake of glucose into cells. This causes a cascade of systemic alterations that may lead to kidney failure, cardiovascular complications, altered tissue healing, retinopathies and gangrene. Diabetes is also associated to increased susceptibility to infections and inflammation.

It has been observed that diabetic patients suffer more often from oral infections such as periodontal disease. Periodontal disease is an infectious-inflammatory disease that leads to destruction of the surrounding tissues of the tooth. It is proposed that the mechanisms responsible for systemic complication are implicated in the development of periodontal disease. This has been evaluated in studies where diabetic patients showed increased levels of inflammatory cytokines, subgingival bacteria and limited response to treatment. Its has also been suggested that established periodontitis in the diabetic patient leads to insulin resistance due to infection and liberation of cytokines from periodontal tissues and thus worsening the diabetic condition.

This study is aimed to establish the response to periodontal treatment with antibiotics and the kinetics of glucose levels in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Must be of legal age (≥18 years old).
* Voluntary participation and signed informed consent.
* Confirmed type I and II diabetes.
* At least 10 teeth present in mouth.

Exclusion Criteria:

* Smokers.
* pregnant women.
* Antibiotic consumption 3 months before inclusion.
* HIV positive or AIDS.
* Allergic reactions to macrolides and specifically to azythromycin.
* Periodontal treatment 6 months before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | 1 year

SECONDARY OUTCOMES:
Bleeding on probing | 1 year
  A sign of gingival inflammation
Clinical attachment level | 1 year
Plaque index | 1 year
Glycemia | 1 year
Probing depth | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Javier E Botero, PhD, Study Director — Universidad de Antioquia, School of dentistry; Fanny L Yepes, DDS, Principal Investigator — Universidad de Antioquia, School of dentistry
Locations (1):
- Universidad de Antioquia, School of dentistry, Medellín, Antioquia, Colombia

REFERENCES:
- [Background] Dandona P, Chaudhuri A, Ghanim H, Mohanty P. Proinflammatory effects of glucose and anti-inflammatory effect of insulin: relevance to cardiovascular disease. Am J Cardiol. 2007 Feb 19;99(4A):15B-26B. doi: 10.1016/j.amjcard.2006.11.003. Epub 2006 Dec 27. PMID 17307055
- [Background] Emrich LJ, Shlossman M, Genco RJ. Periodontal disease in non-insulin-dependent diabetes mellitus. J Periodontol. 1991 Feb;62(2):123-31. doi: 10.1902/jop.1991.62.2.123. PMID 2027060
- [Background] Novak MJ, Potter RM, Blodgett J, Ebersole JL. Periodontal disease in Hispanic Americans with type 2 diabetes. J Periodontol. 2008 Apr;79(4):629-36. doi: 10.1902/jop.2008.070442. PMID 18380555
- [Background] Mealey BL, Rose LF. Diabetes mellitus and inflammatory periodontal diseases. Curr Opin Endocrinol Diabetes Obes. 2008 Apr;15(2):135-41. doi: 10.1097/MED.0b013e3282f824b7. PMID 18316948
- [Background] Ryan ME, Carnu O, Kamer A. The influence of diabetes on the periodontal tissues. J Am Dent Assoc. 2003 Oct;134 Spec No:34S-40S. doi: 10.14219/jada.archive.2003.0370. PMID 18196671
- [Background] Sammalkorpi K. Glucose intolerance in acute infections. J Intern Med. 1989 Jan;225(1):15-9. doi: 10.1111/j.1365-2796.1989.tb00030.x. PMID 2645379
- [Background] Taylor GW, Burt BA, Becker MP, Genco RJ, Shlossman M, Knowler WC, Pettitt DJ. Severe periodontitis and risk for poor glycemic control in patients with non-insulin-dependent diabetes mellitus. J Periodontol. 1996 Oct;67(10 Suppl):1085-93. doi: 10.1902/jop.1996.67.10s.1085. PMID 8910827
- [Background] Garcia R. Periodontal treatment could improve glycaemic control in diabetic patients. Evid Based Dent. 2009;10(1):20-1. doi: 10.1038/sj.ebd.6400633. PMID 19322226
- [Background] Dag A, Firat ET, Arikan S, Kadiroglu AK, Kaplan A. The effect of periodontal therapy on serum TNF-alpha and HbA1c levels in type 2 diabetic patients. Aust Dent J. 2009 Mar;54(1):17-22. doi: 10.1111/j.1834-7819.2008.01083.x. PMID 19228128
- [Background] Madden TE, Herriges B, Boyd LD, Laughlin G, Chiodo G, Rosenstein D. Alterations in HbA1c following minimal or enhanced non-surgical, non-antibiotic treatment of gingivitis or mild periodontitis in type 2 diabetic patients: a pilot trial. J Contemp Dent Pract. 2008 Jul 1;9(5):9-16. PMID 18633464
- [Background] Ernst EJ, Klepser ME, Klepser TB, Nightingale CH, Hunsicker LG. Comparison of the serum and intracellular pharmacokinetics of azithromycin in healthy and diabetic volunteers. Pharmacotherapy. 2000 Jun;20(6):657-61. doi: 10.1592/phco.20.7.657.35176. PMID 10853621